CLINICAL TRIAL: NCT01489683
Title: Effect of Tracheal Lidocaine on Intubating Conditions During Propofol-remifentanil TCI Without Neuromuscular Blockade
Brief Title: Intubating Conditions During Propofol-remifentanil Anesthesia With Topical Lidocaine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Jong Yeop Kim, Associate professor, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AJIRB-MED-CT4-11-073
Record Dates: First submitted 2011-12-07; First posted 2011-12-12 (Estimated); Last update posted 2012-07-16 (Estimated); Status verified 2012-07

CONDITIONS: Drug Usage
Keywords: intubating conditions; propofol; remifentanil; topical lidocaine
MeSH Terms: interventions — Lidocaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- control (Experimental): 3 ml of normal saline was instilled to larynx and trachea
  Interventions: Drug: lidocaine
- lidocaine (Active Comparator): 3 ml of 4% lidocaine was instilled to larynx and trachea before endotracheal intubation
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: lidocaine — 3 ml of 4% lidocaine was instilled to larynx and trachea
  Other Names: 4%lidocaine
  Arms: control
Drug: normal saline — 3 ml of normal saline was instilled to larynx and trachea before endotracheal intubation
  Other Names: control
  Arms: lidocaine

SUMMARY:
When not using neuromuscular blocking agent, even at optimal dosage, target-controlled infusion (TCI) of propofol and remifentanil occasionally produce unsatisfactory intubating conditions. Therefore, the investigators evaluated that the effect of tracheal lidocaine on the intubating conditions for tracheal intubation during anesthesia induction of propofol and remifentanil TCI without neuromuscular blocking agent in day-case anesthesia.

DETAILED DESCRIPTION:
Anesthesia was induced with propofol-remifentanil TCI with the effect-site concentration of 5μg/ml and 5ng/ml, respectively. After TCI, 3 ml of normal saline or 3 ml of 4% lidocaine was instilled to larynx and trachea, following intubation was performed.

ELIGIBILITY:
Inclusion Criteria:

* ASA I, II patients undergoing general anesthesia for reduction of nasal bone fracture

Exclusion Criteria:

* bronchial asthma,
* COPD,
* hypertension,
* anticipated difficult airway

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2011-05; Primary Completion 2012-04 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Overall acceptable conditions for tracheal intubation | baseline from 5 min of TCI was maintained
  Four minutes after start of propofol-remifentanil TCI, 3 ml of normal saline or 3 ml of 4% lidocaine was instilled to larynx and trachea, and one minute later, intubation was performed in double-blinded fashion.

CONTACTS AND LOCATIONS:
Overall Officials: Jong Yeop Kim, MD, Study Director — Ajou University School of Medicine
Locations (1):
- Ajou University School of Medicine, Suwon, South Korea

REFERENCES:
- [Background] Bulow K, Nielsen TG, Lund J. The effect of topical lignocaine on intubating conditions after propofol-alfentanil induction. Acta Anaesthesiol Scand. 1996 Jul;40(6):752-6. doi: 10.1111/j.1399-6576.1996.tb04523.x. PMID 8836274